CLINICAL TRIAL: NCT05072002
Title: Treatment of Low Back Pain in Pregnant Women ; Uses of Drugs and Other Therapies (Acupuncture, Manipulative Medicine, Physical Therapies, Homeopathy) : an Observational Study
Brief Title: Treatment of Low Back Pain in Pregnant Women : Uses of Drugs and Other Therapies
Acronym: LomboMat2021
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI113
Record Dates: First submitted 2021-10-01; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-01

CONDITIONS: Low Back Pain; Pregnancy Related
MeSH Terms: conditions — Low Back Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women with low back pain
  Interventions: Other: no intervention / observational study

INTERVENTIONS:
Other: no intervention / observational study — no intervention / observational study

SUMMARY:
Low back pain is a frequent clinical condition in pregnancy. Drugs treatments are limited. Other therapies are often used, associated or not with drugs (acupuncture, manipulative medicine, physical therapies, homeopathy). Clinical studies suggest a reduction of low back pain with these therapies.

The primary objective of this study is to determinate how many pregnant women use these alternative therapeutics.

In a second time, we want evaluate efficiency of these therapeutics, especially in pain modification and on quality of life.

Our study is a declarative study on pregnant women in Lorraine.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women

Exclusion Criteria:

* medical history of : bifida spina, discal hernia, osteoporosis, vertebral compaction, spondylolisthesis, scoliosis ( over 30°)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women in Lorraine
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of use of other therapies in pregnant women with low back pain ( acunpucture, manipulative medicine, physical therapies, homeopathy) | one day : when each pregnant women submit the questionnaire

SECONDARY OUTCOMES:
Difference of visual analog scale for pain after and before treatment | one day : when each pregnant women submit the questionnaire
Difference of quality life scale after and before treatment | one day : when each pregnant women submit the questionnaire
  Including : affect, walking, sleep, work, social relations. Scale between 0 and 10 for each item

CONTACTS AND LOCATIONS:
Overall Officials: Francis Guillemin, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Centre hospitalier régional universitaire de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No